CLINICAL TRIAL: NCT04900090
Title: Tahiti-families: From Genetic to Phenotype Study of Polynesian Families of Gout Patients
Brief Title: Tahiti-families: Polynesian Families of Gout Patients
Acronym: Tahiti
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Collaborators: Variant Bio, Inc. (Unknown); University of Birmingham (Other); University of San Diego (Other); Ministry of Health, French Polynesia (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC-P00106
Record Dates: First submitted 2021-05-12; First posted 2021-05-25 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Gout
Keywords: Gout; French Polynesia; Epidemiology; Family
MeSH Terms: conditions — Gout | interventions — Epidemiologic Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case group : gout patients (Experimental): Epidemiological study
  Interventions: Other: Epidemiological study
- Control group (Experimental): Epidemiological study
  Interventions: Other: Epidemiological study

INTERVENTIONS:
Other: Epidemiological study — * Clinical phenotypic assessment and neurosensory measures
  * Biological, genetic and metabolomic evaluation
  * Questionnaires (quality of life, gout, life habit, comorbidities)
  * Morphological evaluation by Dual-energy CT scan

SUMMARY:
Gout is a chronic disease caused by the deposit of monosodium urate (MSU) crystals in body tissues secondary to hyperuricemia. Patients with gout suffer severe attacks of acute joint pain. As the disease progresses, the joint pain becomes chronic and associated with disabling and deformative manifestations called tophus. This disease is strongly associated with several comorbidities such as cardiovascular disease and chronic kidney failure. Gout is a very common disease, which is affecting 0.9% of the adult population in France and nearly 4% of the North-American population. Data from New Zealand show a particularly high prevalence of gout among Polynesians (minority populations in New Zealand and other islands of the South Pacific) that would be explained by genetic susceptibility and frequently interrelated metabolic diseases. Data on the Polynesian population in New Caledonia suggest prevalence figures close to 7% and prevalence in French Polynesia is assumed to be higher. International genomic studies of gout and hyperuricaemia have identified alleles associated with the occurrence of gout.

The aim is to focus on families with several gouty members (numerous in French Polynesia, and geographically clustered) in order to enable the study of individuals with monogenic gout or with a low number of variants (= cases) determining in the occurrence of gout, as well as a non-gouty family member (= controls).

Dual-energy CT scan (DECT) allows identification and quantification of UMS crystal deposits in the tissue. The volume of crystals correlates not only with the inflammatory activity of the disease but also with the comorbidities that complicate it. Dual-energy scanning has shown the presence of UMS crystals in some hyperuricemic individuals, which could help to identify those individuals most at risk of developing the disease as they already have the stigma of sub-clinical inflammatory activity.

ELIGIBILITY:
Inclusion Criteria :

Case group :

* Gout patients
* Polynesian origin
* Aged 18 to 80 years
* Agreeing to participate in the study
* Having a 1st or 2nd degree relative who is also gouty and a 1st degree relative of the same generation and sex who is not gouty

Control group :

* Non-gouty individuals who are 1st degree relatives of a gouty patient of the same generation and sex
* Aged 18 to 80 years
* Agreeing to participate in the study

Exclusion Criteria :

* Pregnant women
* Persons under guardianship, curatorship or other legal incapacity
* Persons with a contraindication to Magnetic resonance imaging (MRI) examination
* For non-gouty controls : current hyperuricemic treatment (Allopurinol, Febuxostat, Probenecid or Benzbromarone)
* For gouty case : not participating in the TOPATA study (NCT04812886)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Multiple correlation between genetic variants and clinical presentation | 4 months
  Genome-wide association study (GWAS) aims at identifying genetic variants (genotype) that associated with specific traits (phenotype).
  The link between the genetic variants and the stage of the disease will be sought using a bivariate analysis: Chi-2 tests or Fisher's exact tests in case of small numbers will be implemented

SECONDARY OUTCOMES:
Multiple correlation between disease stage, comorbidities, environmental and metabolomics data | 4 months
  The link between variants will be stablish using a multivariate logistic regression model.- The comorbidities analysed are the following: initial uraemia, glomerular filtration rate (GFR), hypertension, chronic heart failure, diabetes, obesity (BMI > 30), obliterative arterial disease of the lower limbs, history of myocardial infarction, history of cerebrovascular accident
  - The environmental data analysed were as follows: habitus data (alcohol consumption, soft drinks, physical activity)
Multiple correlation between severity of gout, its impact (pain, disease impact, and quality of life), presence of certain genetic variants, metabolomic changes and comorbidities | 4 months
  The link between variants will be stablish using a multivariate logistic regression model. Quality of life will be assessed by the EuroQol questionnaire; perception of hyperuricemia-related illness by the Brief Hyperuricemia Perceptions Questionnaire (BIPQ); body and foot pain in the previous week by a VAS out of 100; activity limitations by the Health Assessment Questionnaire (HAQ-II); foot pain and disability by the Manchester Foot Pain and Disability Index (MFPDI).
Multiple correlation between genetic variants, comorbidities, environmental factors, presence of gout | 4 months
  The link between variants will be stablish using a multivariate logistic regression model. Health status will be assessed by the following elements:
  * Perceived health status: good (modalities "very good" and "good") / bad ("average", "bad" and "very bad")
  * Total number of visits to a health professional in the last 12 monthsThe presence of gout will be determined using a calculation combining and weighting different responses to the questionnaires.
  The diagnosis of gout is retained if the patient meets the 2015 ACR/EULAR criteria for diagnostic classification of gout.

CONTACTS AND LOCATIONS:
Overall Officials: Tristan PASCART, MD PhD, Principal Investigator — GHICL - Hôpital Saint Philibert
Locations (1):
- Centre Hospitalier de Polynésie Française, Papeete, Ville de Pirae, French Polynesia

IPD SHARING:
Plan to Share IPD: No